CLINICAL TRIAL: NCT04911842
Title: Midline Failures: A Comparative, Retrospective Chart Review
Brief Title: Midline Failures: A Comparison Between a Hydrophilic Biomaterial and Thermoplastic Polyurethane
Status: Completed | Type: Observational
Sponsor: Access Vascular Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN 21-001
Record Dates: First submitted 2021-05-25; First posted 2021-06-03 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Midline Catheter

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- TPU: Thermoplastic polyurethane
  Interventions: Device: TPU
- HBM: Hydrophilic BioMaterial
  Interventions: Device: HydroMID

INTERVENTIONS:
Device: HydroMID — Hydrophilic biomaterial
  Groups: HBM
Device: TPU — Thermoplastic polyurethane
  Groups: TPU

SUMMARY:
Retrospective chart review to evaluate and compare the rate of failures between midlines made from different materials

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been inserted with the HydroMID by the vascular access group
* Subjects who have been inserted with a competitor 4 Fr single lumen by the vascular access team

Exclusion Criteria:

* Any off-label use (PICC lines cut to be midlines for any manufacturer)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who needed a 4 Fr single lumen midline
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
The primary objective of this chart review is to evaluate the rates of failure of midlines made from different materials. | retrospective review- March 2021 through May 2021

SECONDARY OUTCOMES:
To compare the proportion of times the midline was used to successfully complete prescribed length. | retrospective review- March 2021 through May 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Joseph Bunch, Romeoville, Illinois, United States